CLINICAL TRIAL: NCT07325383
Title: Evaluating the Safety and Efficacy of N-acetylcysteine Mouthwash on the Prevention of Mucositis in Patients Undergoing Hematopoietic Stem Cell Transplantation: a Double-blind Randomized Clinical Trial
Brief Title: Safety and Efficacy of N-Acetylcysteine Mouthwash in Prevention of Mucositis in HSCT Patients
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Tehran University of Medical Sciences (Other)
Collaborators: Research Institute for Oncology- Hematology and Cell Therapy (RIOHCT), Tehran University of Medical Sciences, Iran (Unknown)
Responsible Party: Principal Investigator, Bita Shahrami, PharmD, iBCPS, FCCP Assistant; Professor at Tehran University of Medical Sciences (TUMS), Tehran University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: IR.TUMS.DENTISTRY.REC.1403.048; IRCT20140818018842N42 (Registry Identifier: Iranian Registry of Clinical Trials)
Record Dates: First submitted 2025-11-16; First posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Oral Mucositis; Hematopoietic Stem Cell Transplantation (HSCT)
Keywords: N-Acetylcysteine; Oral Mucositis; Hematopoietic Stem Cell Transplantation; Chemotherapy-Induced Mucositis; Mouthwash
MeSH Terms: conditions — Stomatitis | interventions — Acetylcysteine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- N-Acetylcysteine group (Experimental): Participants in this group receive 2400 mg of N-acetylcysteine daily as an oral mouthwash, divided into four doses per day. The intervention starts at the beginning of the conditioning regimen and continues until day 14 after hematopoietic stem cell transplantation.
  Interventions: Drug: N-Acetylcysteine 600mg/tab
- Placebo group (Placebo Comparator): Participants in this group receive a placebo mouthwash with identical appearance, taste, and administration schedule as the NAC mouthwash. The placebo contains no active pharmaceutical ingredients and is administered four times daily from the start of conditioning until day 14 post-transplantation.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: N-Acetylcysteine 600mg/tab — Each dose consists of one 600 mg effervescent tablet of N-acetylcysteine (NAC) dissolved in 20 mL of sodium carbonate solution. Participants receive this mouthwash four times daily, totaling 2400 mg of NAC per day. The solution is used as an oral rinse (swish and spit) and is not intended to be swallowed. Administration begins with the conditioning regimen and continues until day 14 after HSCT.
  Other Names: NAC
  Arms: N-Acetylcysteine group
Drug: Placebo — Each dose consists of one placebo effervescent tablet, identical in appearance and packaging to the N-acetylcysteine tablets, dissolved in 20 mL of sodium carbonate solution. Participants use this placebo mouthwash four times daily as an oral rinse (swish and spit), starting from the conditioning regimen and continuing until day 14 post-transplantation. The placebo contains no active pharmaceutical ingredients.
  Arms: Placebo group

SUMMARY:
Oral mucositis (OM) is one of the most frequent complications in patients who undergo HSCT. It not only causes severe discomfort but also affects treatment adherence and increases hospital stays. In this study, we aim to assess whether using N-acetylcysteine mouthwash can safely and effectively prevent OM. The trial is randomized and conducted in the hematology wards of TUMS-affiliated RIOHCT, including both autologous and allogeneic HSCT patients.

DETAILED DESCRIPTION:
This randomized, double-blind, placebo-controlled clinical trial evaluates the safety and efficacy of N-acetylcysteine (NAC) mouthwash in preventing oral mucositis (OM) in patients undergoing hematopoietic stem cell transplantation (HSCT). Oral mucositis is one of the most common and severe complications following HSCT, significantly affecting patient quality of life, treatment adherence, and duration of hospitalization.

A total of 100 patients undergoing autologous or allogeneic HSCT were enrolled and randomly assigned into two parallel groups: an intervention group and a placebo group. The intervention group received 2400 mg of N-acetylcysteine daily as a mouthwash, while the control group received a placebo mouthwash with identical appearance and administration protocol. Both patients and healthcare providers were blinded to group allocation.

The study was conducted at the Research Institute of Oncology, Hematology, and Cell Therapy (RIOHCT), located in Shariati Hospital and affiliated with Tehran University of Medical Sciences. Daily evaluations for the incidence and severity of mucositis were performed using the World Health Organization (WHO) mucositis grading scale.

The primary objective is to assess the efficacy of prophylactic NAC mouthwash in reducing the incidence and severity of OM, particularly grades 3 and 4. Secondary objectives include examining the effect of NAC mouthwash on hospitalization length after engraftment and determining the safety profile of the intervention. Findings from this study may support the introduction of NAC mouthwash as a preventive strategy against mucositis in HSCT patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing hematopoietic stem cell transplantation (HSCT), including both allogeneic and autologous transplants
* Age ≥18 years
* Ability to provide informed consent

Exclusion Criteria:

* Known hypersensitivity to N-acetylcysteine or any components of the effervescent tablets
* Inability to adhere to the proper use of mouthwash
* Systemic use of N-acetylcysteine during the study period
* Pregnancy or lactation

Ages: 18 Years to 66 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2024-08-18 (Actual); Primary Completion 2025-03-08 (Actual); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Incidence of oral mucositis | From day 1 of conditioning to day +14 post-transplantation.
  Oral mucositis is a painful and debilitating complication of hematopoietic stem cell transplantation, characterized by erythema, edema, and ulcerations of the oral mucosa. The incidence of mucositis is assessed daily from the beginning of the conditioning regimen until day +14 post-transplantation. The World Health Organization (WHO) Oral Toxicity Scale is used to grade the severity of mucositis. The presence of grade ≥1 mucositis is recorded as incidence.
Incidence of N-acetylcysteine-related Adverse Events | Clinical examination is performed daily from the beginning of the conditioning regimen until day +14 post-transplantation.
  Participants are monitored daily for any adverse events potentially related to the use of N-acetylcysteine mouthwash. Adverse events include non-immune anaphylaxis reactions, cardiovascular reactions, dermatologic reactions (such as rash or pruritus), and gastrointestinal reactions (such as nausea or vomiting).
Incidence of Severe Oral Mucositis | From day 1 of conditioning to day +14 post-transplantation
  Severe oral mucositis is defined as grade 3 or 4 according to the World Health Organization (WHO) Oral Toxicity Scale. Participants are assessed daily to determine the presence and severity of mucositis. The incidence of severe mucositis (grade ≥3) is recorded during the study period.

SECONDARY OUTCOMES:
Length of Hospitalization | From hospital admission through hospital discharge, up to Day +60 post-transplantation
  The number of days from admission for hematopoietic stem cell transplantation until hospital discharge. Data are obtained from the patients' medical records. This outcome reflects overall clinical recovery and is used to evaluate the potential supportive effect of N-acetylcysteine on hospitalization duration.

CONTACTS AND LOCATIONS:
Locations (1):
- Research Institute of Oncology, Hematology, and Cell Therapy, Shariati Hospital, Tehran, Iran

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Moslehi A, Taghizadeh-Ghehi M, Gholami K, Hadjibabaie M, Jahangard-Rafsanjani Z, Sarayani A, Javadi M, Esfandbod M, Ghavamzadeh A. N-acetyl cysteine for prevention of oral mucositis in hematopoietic SCT: a double-blind, randomized, placebo-controlled trial. Bone Marrow Transplant. 2014 Jun;49(6):818-23. doi: 10.1038/bmt.2014.34. Epub 2014 Mar 10. PMID 24614837